CLINICAL TRIAL: NCT03185949
Title: Efficacy and Safety of EndoBar Bariatric Embolization for Weight Management in People With Obesity
Brief Title: The Lowering Weight in Severe Obesity by Embolization of the Gastric Artery Trial
Acronym: LOSEIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endobar Solutions LLC (Industry)
Collaborators: OB KLINIKA a.s. Pod Krejcárkem 975 Praha 3 - Žižkov Tel.: +420 255 725 110 (Unknown); Na Homolce Hospital (Other); High Tech Med Consult (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ESC-14-001
Record Dates: First submitted 2017-05-09; First posted 2017-06-14 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Embolization; Left Gastric Artery
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: This study is a prospective, sham controlled, single-blind 12-month trial with 1:1 randomization. A maximum of 40 subjects (obese men and women who have a body mass index (BMI) of 35.0-50.0 kg/m2) will be enrolled in the study. Eligible subjects will be randomized to treatment with Endobar Therapy (n = 20) or sham procedure control (n = 20). Endobar Therapy involves catheter-based embolization of the left gastric artery. All subjects in both Endobar Therapy and Sham Control groups will receive Lifestyle Therapy (behavioral and diet education). At the end of 6 months all subjects randomized to the Sham Control group will receive catheter-based embolization of the left gastric artery. Both Endobar Therapy and Sham Control crossover to Endobar Therapy groups will be followed for a total of 12 months
Who Masked: Participant, Outcomes Assessor
Masking Description: * Interventional Group: These subjects will undergo catheter-based embolization.
  * Sham Control Group: These subjects will not undergo femoral artery catheterization. Instead, lidocaine will be injected subcutaneously at the femoral artery site in the Sham Control group. Since all patients will have received at least sedation, they will not be aware of what has been done, and thus be blind to their treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Sedation and subcutaneous lidocaine (Sham Comparator): Lidocaine injected at the femoral artery site. This patients will undergo behavioral therapy for 6 months and will crossover and will receive bariatric embolization.
  Interventions: Device: Endobar Infusion Catheter System; Behavioral: Behavioral therapy
- interventional: bariatric embolization (Experimental): • In patients randomized to intervention bariatric embolization will be performed using Endobar Infusion Catheter System. After procedure patients will undergo behavioral therapy
  Interventions: Device: Endobar Infusion Catheter System; Behavioral: Behavioral therapy

INTERVENTIONS:
Device: Endobar Infusion Catheter System — Bariatric embolization with microspheres using Endobar Infusion Catheter System
Behavioral: Behavioral therapy — Healthy diet and exercise

SUMMARY:
To evaluate the efficacy and safety of the Endobar gastric embolization system for the treatment of obesity before continuing to a larger Pivotal Trial.

Investigational Device The investigational device in this clinical study is the Endobar Infusion Catheter System - a disposable system consisting of an occlusion balloon catheter, a Smart Manifold delivery system.

Study Design/Planned Number of Subjects This study is a prospective, sham controlled, single-blind 12-month trial with 1:1 randomization. A maximum of 40 subjects (obese men and women who have a body mass index (BMI) of 35.0-50.0 kg/m2) will be enrolled in the study. Eligible subjects will be randomized to treatment with Endobar Therapy (n = 20) or sham procedure control (n = 20). Endobar Therapy involves catheter-based embolization of the left gastric artery. All subjects in both Endobar Therapy and Sham Control groups will receive Lifestyle Therapy (behavioral and diet education). At the end of 6 months all subjects randomized to the Sham Control group will receive catheter-based embolization of the left gastric artery. Both Endobar Therapy and Sham Control crossover to Endobar Therapy groups will be followed for a total of 12 months.

Study Duration The duration of the study is expected to last approximately 18 months from the first enrollment . An additional 12 months to the study closeout after the last follow-up.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Objective The objective of this study is to conduct a sham controlled randomized trial to evaluate the efficacy and safety of the Endobar System for the treatment of obesity. Efficacy, Safety, and secondary outcomes will be evaluated at 6 and 12 months to allow expansion of the investigation into a larger, pivotal clinical study.

Study Design This is a prospective randomized, single blind, active treatment and sham controlled, single-center trial . After the informed consent and screening process are completed, all subjects who are eligible and wish to participate in the study will undergo baseline testing. Those who complete baseline testing will be randomized to either Endobar Therapy (ET) or Sham Treatment (ST) for 52 weeks. Both groups will be given lifestyle therapy for weight loss, which involves treatment with a behavioral education weight loss program delivered as 19 individual sessions in person over 52 weeks. Endobar Therapy involves catheter-based embolization of the left gastric artery. After 26 weeks, the ET group will continue to be monitored for an addition 26 weeks and the ST subjects will be given ET and monitored for 26 weeks. The duration of the entire study will be 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • BMI 35.0-50.0 kg/m2 at time of screening

  * Women of childbearing potential must agree to use at least one form of birth control (prescription hormonal contraceptives, diaphragm, IUD, condoms with or without spermicide, or voluntary abstinence) from time of study enrollment through study exit.
  * Willing and able to provide informed consent

Exclusion Criteria:

* • Previous bariatric, gastric pancreatic, hepatic, and/or splenic surgery

  * History of duodenal or gastric ulcers or regularly taking medications (therapy >1 day per week) that can cause ulcers (e.g., non-steroidal anti-inflammatory drugs)
  * Prior radiation to the upper abdomen
  * Prior embolization to the stomach, spleen or liver
  * Portal venous hypertension
  * Active H. pylori infection
  * Uncontrolled hypertension (> 160/100 with or without medication).
  * Diabetes (determined by medical history, fasting blood glucose or results of an oral glucose tolerance test)
  * Serum triglyceride > 400 mg/dL at screening.
  * Class 4 or 5 surgical risk based on standard ASA criteria (Saklad M. Grading of patients for surgical procedures. Anesthesiol. 1941; 2:281-4).
  * Severe pulmonary or cardiovascular disease defined as a history or evidence of serious cardiovascular disease, including myocardial infarction, acute coronary syndrome, coronary revascularization, heart failure requiring medications, history of sudden cardiac death, or NYHA (New York Heart Association) class III or IV heart failure (defined below):

    * Class III: patients with marked limitation of activity; they are comfortable only at rest.
    * Class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest.
  * Coagulation disorders (platelets < 100,000, PT > 2 seconds above control or INR > 1.5 at screening).
  * Anemia (Hb < 10.0 g/dL) at screening.
  * Malignancy in the last 5 years (except for non-melanoma skin cancer).
  * Evidence of other significant organ system dysfunction (e.g. cirrhosis, renal failure)
  * Pregnant or lactating.
  * History of substance abuse in last 3 years.
  * Thyroid Stimulating Hormone (TSH) >2.0 x upper limit of normal at screening.
  * Taking prescription or over-the-counter medications for weight loss in the last 3 months before screening, or planning to participate in a commercial weight loss program in the next 5 years.
  * Taking diuretic medication for congestive heart failure or edema.
  * Evidence of significant mucosal inflammation, ulceration or ischemia detected on endoscopy, and those with unsuitable left gastric anatomy as judged by the study site physician will be excluded
  * Psychiatric illness that could affect compliance with the study, as judged by the site principle investigator.
  * Unable to complete screening requirements (compliance with visits and dietary record)
  * Taking medication once or more per week that causes weight gain (e.g. atypical antipsychotics, monoamine oxidase inhibitors, lithium, selected anticonvulsants, tamoxifen, glucocorticoids)
  * Chronic abdominal pain that would potentially complicate management.
  * Unstable weight (>3% change; self-reported) over the previous 2 months at time of screening.
  * Subjects whom the site investigator, research team, or the study medical monitor feel is not able to participate in the study for any reason, including poor general health or unable/unwilling to follow the study protocol.

Ages: 21 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fried, MD, Principal Investigator — OB klinika a.s., Prague, Czech Republic; Peter Neuzil, MD, Principal Investigator — Na Homolce Hospital, Prague, Czech Republic; Vivek Reddy, MD, Principal Investigator — Mount Sinai Medical Center, New York, NY, USA
Locations (1):
- OB klinika a.s., Pod Krejcárkem 975, Praha 3 - Žižkov, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Neuzil P, Musikantow D, Sramkova P, Rosen R, Kipshidze N, Kipshidze N, Fried M. Transcatheter Bariatric Embolotherapy for Weight Reduction in Obesity. J Am Coll Cardiol. 2020 Nov 17;76(20):2305-2317. doi: 10.1016/j.jacc.2020.09.550. PMID 33183504

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Control: Lidocaine injected at the femoral artery site. This patients will undergo behavioral therapy for 6 months and will crossover and will receive bariatric embolization.
  Endobar Infusion Catheter System: Bariatric embolization with microspheres using Endobar Infusion Catheter System
  Behavioral therapy: Healthy diet and exercise
- Percutaneous Transcatheter Embolotherapy: In patients randomized to intervention bariatric embolization will be performed using Endobar Infusion Catheter System. After procedure patients will undergo behavioral therapy
  Endobar Infusion Catheter System: Bariatric embolization with microspheres using Endobar Infusion Catheter System
  Behavioral therapy: Healthy diet and exercise
Period: ITT Analysis
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Started (Assessed for eligibility) | 22 | 22
Completed | 18 | 19
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3
Period: PP Analysis
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Started (All participants who were part of the ITT Population) | 18 | 19
Completed | 16 | 15
Not Completed | 2 | 4
Not completed — Protocol Violation | 2 | 2
Not completed — Failed/Incomplete LGA embolization | 0 | 2
Period: Cross-over at 6 Months
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Started (At 6 months, study participants were unblinded and those in the sham control group were given the option to cross over.) | 16 | 0
Completed | 15 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Percutaneous Transcathether Embolotherapy: In patients randomized to intervention bariatric embolization will be performed using Endobar Infusion Catheter System. After procedure patients will undergo behavioral therapy
  Endobar Infusion Catheter System: Bariatric embolization with microspheres using Endobar Infusion Catheter System
  Behavioral therapy: Healthy diet and exercise
- Total: Total of all reporting groups
Arm/Group | Sham Control | Percutaneous Transcathether Embolotherapy | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (9.4) | 46.4 (10.3) | 45.55 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 1 | 7 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 22 | 22 | 44
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 38.93 (3.8) | 40.2 (3.7) | 39.58 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: 1. Difference in percent total body weight (% TBWL) loss at 6 months between the Sham Control and Endobar Therapy groups. This is calculated as the difference in body weight from baseline to 6 months, relative to the baseline weight (i.e, initial weight - 6 month weight / initial weight) x 100%). The mean (i.e., average) total body weight loss of both groups was compared to assess whether there was a meaningful difference.
  2. Percent total body weight loss (%TBWL) at 12 months in the group randomized to the initial Endobar Therapy alone. This is calculated as the difference in body weight from baseline to 12 months, relative to the baseline weight (i.e, initial weight - 12 month weight / initial weight) x 100%).
Time Frame: 1) 6 months post-procedure/sham and 2) 12 months post-procedure
Population: The ITT is representative of all randomized subjects who underwent either the sham or PTE, regardless of follow-up compliance. The PP represents subjects treated and compliant to study treatment and follow-up visits per the protocol, no major protocol deviations, or protocol violations. Note for 12 months post-procedure, only those initially randomized to PTE were followed for 12 months. The sham control, pursuant to the study protocol, were only followed for 6 months post-procedure.
Measure: Mean (95% Confidence Interval); unit: Percent change
Groups:
- Percutaneous Transcatheter Embolotherapy: • In patients randomized to intervention bariatric embolization will be performed using Endobar Infusion Catheter System. After procedure patients will undergo behavioral therapy
  Endobar Infusion Catheter System: Bariatric embolization with microspheres using Endobar Infusion Catheter System
  Behavioral therapy: Healthy diet and exercise
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 18 | 19
Percent change
  6 Months: ITT Population | 2.8 [0.9 to 4.7] | 6.4 [3.2 to 9.6]
  6 Months: PP Population: number analyzed (Participants) | 16 | 15
  6 Months: PP Population | 1.8 [0.5 to 3.0] | 8.3 [4.9 to 11.6]
  12 Months: ITT Population: number analyzed (Participants) | 0 | 19
  12 Months: ITT Population |  | 6.5 [3.0 to 10.0]
  12 Months: PP Population: number analyzed (Participants) | 0 | 15
  12 Months: PP Population |  | 9.3 [5.3 to 13.3]

2. Primary Outcome: Number of Patients With Adverse Events
Description: The Incidence of device-, procedure- and therapy-related adverse events up to 12 months post-procedure.
Time Frame: 12 months post-randomization
Population: Safety Population (i.e. any participant who consented to be in the study and underwent either the sham or therapy procedure). Each count indicates a participant who reported experiencing the described event.
Measure: Number; unit: participants
Groups:
- Percutaneous Transcatheter Embolotherapy: Includes those initially randomized to the therapy group at screening + those who crossed over at 6 months when randomization was unblinded.
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 20 | 34
participants
  Asymptomatic Ulcers | 0 | 5
  Epigastring Pain | 3 | 4
  Epigastric Pressure | 0 | 3
  Nausea | 4 | 7
  Vomitting | 5 | 7

3. Primary Outcome: Absolute Weight Loss (kg)
Description: 6-month change: The absolute difference in the initial and 6-month weight (kg) (i.e., initial - 6 month weight). These changes were averaged for each group and compared between the two groups to assess whether there was a meaningful difference.
  12-month change: The absolute difference in the initial and 12-month weight (kg) (i.e., initial - 12 month weight).
Time Frame: 6 months post-procedure/sham and 12 months post-procedure
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kilograms
Groups:
- Percutaneous Transcatheter Embolotherapy: Bariatric embolization will be performed using Endobar Infusion Catheter System. After the procedure, patients will undergo behavioral therapy.
  Endobar Infusion Catheter System: Bariatric embolization with microspheres using Endobar Infusion Catheter System
  Behavioral therapy: Healthy diet and exercise
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 18 | 19
kilograms
  6 Months: ITT Population | 3.0 [0.9 to 5.0] | 7.4 [3.8 to 11.0]
  6 Months: PP Population: number analyzed (Participants) | 16 | 15
  6 Months: PP Population | 9.4 [5.6 to 13.2] | 1.9 [0.5 to 3.3]
  12 Months: ITT: number analyzed (Participants) | 0 | 19
  12 Months: ITT |  | 7.8 [3.6 to 12.0]
  12 Months: PP: number analyzed (Participants) | 0 | 15
  12 Months: PP |  | 9.3 [4.9 to 13.8]

4. Secondary Outcome: Percent Excess Body Weight (%EBWL) Loss
Description: Percent excess body weight loss (% EBWL) is calculated by dividing the absolute weight loss divided by baseline excess weight and multiplying by 100% (i.e., excess weight / initial weight x 100%). Excess weight is defined as the difference between current weight and ideal weight.
  %EBWL was calculated for the following time points:
  1. 6 months: absolute weight loss was the difference from baseline to 6 months. %EBWL was averaged for each group and compared to assess whether there was a meaningful difference between the groups.
  2. 12 months: absolute weight loss was the difference from baseline to 12 months.
  Note, excess weight was determined from ideal body weights based on a BMI=25 kg/m2.
Time Frame: 1) 6 months post-procedure/sham and 2) 12 months post-procedure
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: EBWL %
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 18 | 19
EBWL %
  6 Months: ITT Population | 8.6 [2.5 to 14.7] | 17.1 [8.5 to 25.7]
  6 Months: PP Population: number analyzed (Participants) | 16 | 15
  6 Months: PP Population | 5.4 [1.7 to 9.1] | 22.3 [13.4 to 31.1]
  12 Months: ITT Population: number analyzed (Participants) | 0 | 19
  12 Months: ITT Population |  | 17.3 [7.9 to 26.8]
  12 Months: PP Population: number analyzed (Participants) | 0 | 15
  12 Months: PP Population |  | 21.8 [11.1 to 32.4]

5. Secondary Outcome: Number of Patients With Weight Loss ≥5%
Description: Proportion of subjects who achieve ≥5% total body weight loss from baseline vs. those who do not
Time Frame: 6 months post-procedure/sham
Population: The intention-to-treat (ITT) and per-protocol (PP) groups. The ITT population is representative of all randomized subjects who underwent either the sham or the therapeutic procedure, regardless of when they withdrew from the study or not post-procedure. The PP population represents subjects treated and complaint to study treatment and follow-up visits per the protocol, no major protocol deviations, or protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 18 | 19
Participants
  ITT Population: < 5% | 14 | 10
  ITT Population: ≥ 5% | 4 | 9
  PP Population: number analyzed (Participants) | 16 | 15
  PP Population: < 5% | 14 | 6
  PP Population: ≥ 5% | 2 | 9

6. Secondary Outcome: 6 Month Change in Lipids
Description: 6-month change (from baseline) in lipids for both groups. Unit of Measure: mg/dL
Time Frame: 6 months post-procedure/sham
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 18 | 19
mmol/L
  Total Cholesterol - Baseline | 5.23 (0.81) | 4.69 (0.71)
  Total Cholesterol - 6 Months | 4.99 (0.70) | 4.94 (0.71)
  Low-Density Lipoprotein (LDL) - Baseline | 1.23 (0.74) | 1.29 (0.69)
  Low-Density Lipoprotein (LDL) - 6 Months | 1.26 (0.64) | 1.28 (0.68)
  High-Density Lipoprotein (HDL) - Baseline | 1.23 (0.28) | 1.29 (0.32)
  High-Density Lipoprotein (HDL) - 6 Months | 1.26 (0.21) | 1.28 (0.26)
  Triglyceride - Baseline | 1.29 (0.52) | 1.34 (0.76)
  Triglyceride - 6 Months | 1.41 (0.74) | 1.40 (1.14)

7. Secondary Outcome: 6 and 12 Month Change in Blood Pressure
Description: Change in absolute blood pressure levels from baseline to 6 months for both groups and baseline to 12 months for the initial treatment group.
  Unit of Measure: mmHg
Time Frame: 6 months post-procedure/sham and 12 months post-procedure
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
Number analyzed (Participants) | 18 | 19
mmHg
  6 Months: Systolic Blood Pressure | -3.7 [-13.6 to 6.2] | 2.3 [-5.0 to 9.7]
  6 Months: Diastolic Blood Pressure | -0.6 [-6.6 to 5.5] | 2.8 [-0.3 to 5.9]
  12 Months: Systolic Blood Pressure: number analyzed (Participants) | 0 | 19
  12 Months: Systolic Blood Pressure |  | -1.8 [-8.6 to 4.9]
  12 Months: Diastolic Blood Pressure: number analyzed (Participants) | 0 | 19
  12 Months: Diastolic Blood Pressure |  | -9.7 [-17.7 to -1.7]

8. Other Pre Specified Outcome: Ghrelin Levels
Description: Unit of Measure: pg/mL
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Glucagon-like Peptide 1 Concentrations
Description: Changes in Glucagon-like peptide 1 concentrations Unit of Measure: pg/mL
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Oral Glucose Tolerance and Insulin Sensitivity
Description: Changes in OGTT and Insulin Sensitivity Unit of measure:milligrams/deciliter (mg/dL)
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Insulin Sensitivity
Description: Unit of measure: mg/min
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in Mood (Depression/Anxiety)
Description: Unit of Measure: Beck Depression Index
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Quality-of-life
Description: Change in the subdomains and overall Quality of Life Unit of Measure: IWQOL
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Eating Behavior
Description: Unit of Measure: Eating Questionnaire Scores
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Volume of Meal Test Consumed to Achieve Satiation: Satiation Drink Test.
Description: Change in satiety and other parameters associated with this test Unit of Measure: numerical scale from 0-5
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Results From Endoscopy
Description: Photos and clinical reports analyzed
Time Frame: 12 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Gastric Motility/Emptying
Description: Unit of Measure: (t 1/2) in minutes
Time Frame: [Time Frame: 6-12 months]
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1) 12 Months for those initially randomized to PTE (therapy group); 2) 6 months for those initially randomized to sham group; 3) 6 months for those who crossed over to PTE (therapy group) after unblinding point of the study, pursuant to the study protocol.
Groups:
- Sham Control: Those who were initially randomized to the sham control group and followed up for 6 months post-sham.
- Percutaneous Transcatheter Embolotherapy: Those initially randomized to PTE and those who crossed over to PTE at 6 months post-sham during unblinding of the study.
Arm/Group | Sham Control | Percutaneous Transcatheter Embolotherapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/34
Other Adverse Events (participants affected / at risk) | 0/20 | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Control (N=20) | Percutaneous Transcatheter Embolotherapy (N=34)
Chronic high-grade atherosclerotic stenosis of the external iliac artery (Vascular disorders) | 0 | 1 — Patient with previously unrecognized chronic high-grade atherosclerotic stenosis of the external iliac artery underwent surgical correction. The SAE was determined to not be related to the device or procedure by the site investigator.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Control (N=20) | Percutaneous Transcatheter Embolotherapy (N=34)
Asymptomatic Ulceration (Gastrointestinal disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03185949/Prot_SAP_000.pdf